CLINICAL TRIAL: NCT03358264
Title: Effect of L-Citrulline Supplementation on Arginase Activity and Vascular Function in Type II Diabetes Mellitus
Brief Title: Effect of L-Citrulline Supplementation on Arginase Activity and Vascular Function in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia Shatanawi, Associate Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pharmacology-Medicine-UJ
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Vascular dysfunction, L-citrulline, arginase
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetic patients (Experimental): L-citrulline at a dose of 2000 mg per day for a period of 1 month will be administered to type 2 diabetic patients with HbA1c>6
  Interventions: Dietary Supplement: L-citrulline
- Healthy volunteers (Experimental): L-citrulline at a dose of 2000 mg per day for a period of 1 month will be administered to non-diabetic healthy volunteers
  Interventions: Dietary Supplement: L-citrulline

INTERVENTIONS:
Dietary Supplement: L-citrulline — Amino acid supplement

SUMMARY:
Arginase has recently been implicated in an array of vascular conditions including atherosclerosis , hypertension and vascular complication of diabetes. In this study we will determine of L-citrulline; a natural amino acid that is known to have inhibitory effects on arginase activity, on vascular function in type 2 diabetic patients.

DETAILED DESCRIPTION:
Vascular dysfunction is a major cause of morbidity and mortality in diabetic patients. The pathological process is characterized by impaired endothelial cell production of the vasodilator and antiplatelet adhesion factor nitric oxide (NO) and/or decreased NO bioavailability. NO is a major regulator of vascular tone and integrity. In endothelial cells, NO is produced by activity of endothelial NO synthase (eNOS) on its substrate L-arginine. Reduced availability of L-arginine to eNOS has been implicated in vascular dysfunction in diabetes and a variety of other disease conditions. Arginase, which metabolizes L-arginine to urea and ornithine, competes directly with NOS for L-arginine. Hence increases in arginase activity can decrease tissue and cellular arginine levels, reducing its availability to eNOS and decreasing No production. During diabetes, elevated levels of arginase can compete with NOS for available arginine thus reducing vascular NO. We have recently shown that arginase activity is elevated in diabetes. In this proposal we implement a method of flow mediate dilation (FMD) to assess vascular function in diabetic patients. We will study the relation of our vascular function findings with arginase activity levels. We propose that arginase activity measurements could be novel marker of vascular dysfunction in diabetes. The effect of the natural amino acid supplements (L-citrulline) on levels of arginase activity in diabetic patients and vascular function will also be studied.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes Diabetic state: HbA1c>6

Exclusion Criteria:

-

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
arginase activity | 1 month
  Levels of arginase activity enzyme will be measured in plasma in subjects before and after l-citrulline supplementation
Vascular function | 1 month
  forearm vascular function will be assessed by flow mediated dilation of brachial blood vessels before and after L-citrulline supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shatanawi A, Momani, MS. Plasma arginase activity is elevated in type 2 diabetic patients. Biomedical Research-India 28(9): 4102-4106, 2017